CLINICAL TRIAL: NCT06102278
Title: Machine Learning Models for Predicting Postoperative Peritoneal Metastasis After Hepatocellular Carcinoma Rupture
Brief Title: ML Models for Predicting Postoperative Peritoneal Metastasis After Hepatocellular Carcinoma Rupture
Status: Completed | Type: Observational
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: PM-01
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Peritoneal Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: All cases were randomly grouped according to 7:3, with 70% defined as the training group
  Interventions: Other: Peritoneal Metastasis
- Validation cohort: All cases were randomly grouped according to 7:3, with 30% defined as the validation group
  Interventions: Other: Peritoneal Metastasis

INTERVENTIONS:
Other: Peritoneal Metastasis — Patients experiencing postoperative peritoneal metastasis

SUMMARY:
This study aimed to address the issue of peritoneal metastasis (PM) following the rupture of hepatocellular carcinoma (HCC) and its adverse impact on patient prognosis. Clinical data from 522 patients with ruptured HCC who underwent surgery at seven different medical centers were collected and analyzed. Machine learning models were employed for analysis and prediction.

ELIGIBILITY:
Inclusion Criteria:(1) HCC confirmed by pathologists (2) two preoperative imaging findings suggestive of tumor rupture (3) R0 resection (4) first tumor detection -

Exclusion Criteria:(1) previous antitumor therapy (2) combination of other types of tumors (3) incomplete clinical data

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 522 rHCC patients who underwent radical hepatectomy
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 2018-2023
  Overall survival (OS) was defined as the time from the date of surgery to death

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided